CLINICAL TRIAL: NCT03122639
Title: Vascular Endothelial Activation in Obstructive Sleep Apnea
Brief Title: Endothelial Function in Obstructive Sleep Apnea
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Sanja Jelic, Associate Professor, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: AAAR0444; 2R01HL106041-06A1 (NIH)
Record Dates: First submitted 2017-04-12; First posted 2017-04-21 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Obstructive Sleep Apnea of Adult
MeSH Terms: interventions — Atorvastatin; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Intervention Model Description: Randomized double blind design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Active drug and placebo will be made identical in appearance and given to participants in a blinded fashion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Active Comparator): OSA patients who adhered or did not adhere with CPAP will be randomized 1:1 to treatment (atorvastatin 10 mg daily) or control group (placebo).
  Interventions: Drug: Atorvastatin 10mg
- Control (Placebo Comparator): OSA patients who adhered or did not adhere with CPAP will be randomized 1:1 to treatment (atorvastatin 10 mg daily) or control group (placebo).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin 10mg — Atorvastatin 10 mg daily for 28 days will be randomly allocated to OSA patients regardless of adherence with CPAP. CPAP is a standard of care for OSA and will be prescribed by care providers not associated with this study based on clinical indications. The investigators will have no role in prescribing CPAP. Atorvastatin and placebo will be encapsulated to appear identical and dispensed by the research pharmacy.
  Other Names: statin
  Arms: Treatment
Drug: Placebo — Placebo daily for 28 days will be randomly allocated to OSA patients regardless of adherence with CPAP. CPAP is a standard of care for OSA and will be prescribed by care providers not associated with this study based on clinical indications. The investigators will have no role in prescribing CPAP. Atorvastatin and placebo will be encapsulated to appear identical and dispensed by the research pharmacy.
  Arms: Control

SUMMARY:
Obstructive sleep apnea (OSA), a condition that affects a quarter of the Western adults, triples the risk for cardiovascular diseases and increases all-cause mortality. Intermittent hypoxia (IH) during transient cessation of breathing in OSA leads to endothelial inflammation, a key step in the initiation and progression of cardiovascular disease. However, the mechanisms that mediate IH-induced endothelial inflammation remain unclear and, consequently, no targeted therapy is available for vascular manifestations of OSA. Using endothelial cells (ECs) freshly harvested from OSA patients, they study team has identified impaired complement inhibition as an initial stimulus for endothelial inflammation in IH, thereby linking for the first time complement activation to vascular risk in OSA. The investigators found that a major complement inhibitor cluster of differentiation (CD59), a plasma membrane protein that inhibits the formation of the terminal complement membrane attack complex (MAC) and protects host cells from complement injury, is internalized from the EC surface in OSA patients. Consequent MAC deposition initiates endothelial inflammation in IH. Importantly, the investigators showed that IH does not significantly affect inflammation in ECs in the absence of complement, suggesting that complement activation has an essential role in endothelial inflammation in OSA. Interestingly, internalization of CD59 in IH appears to be cholesterol-dependent and statins prevent MAC deposition on ECs in IH in a CD59-dependent manner, suggesting a novel therapeutic strategy to reduce vascular risk in OSA. This led the study team to hypothesize that IH-induced cellular cholesterol accumulation reduces complement inhibition via increased internalization of CD59 from the EC surface leading to increased MAC deposition, and that treatment of OSA with continuous positive airway pressure (CPAP) and/or statins reverses endothelial dysfunction by restoring complement inhibition.

DETAILED DESCRIPTION:
To address the hypothesis, the investigators seek to determine whether statins prevent endothelial dysfunction in OSA by restoring complement inhibition. The preliminary data indicate that the expression of CD59 on the EC surface is preserved in OSA patients who are receiving statins and that statins prevent CD59 internalization and MAC deposition in IH leading to reduced inflammation. The study proposes to determine whether statins restore endothelial protection against complement activity in OSA patients using double-blind placebo-controlled parallel group randomized study design. The hypothesis: The proportion of CD59 on the EC surface is increased while MAC deposition is decreased after 4 weeks of atorvastatin 10 mg daily compared with placebo in OSA patients who adhere with CPAP or do not adhere with CPAP.

The proposed studies may advance our understanding of vascular dysfunction in OSA and provide the basis for large, long-term clinical trials of novel therapeutic strategies, such as addition of statins to the standard CPAP therapy, for preventing and/or reversing vascular risk in OSA.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years with newly diagnosed obstructive sleep apnea (OSA) who were never treated with CPAP. OSA is defined as apnea-hypopnea index (AHI) ≥5 events/hour of sleep.

Exclusion Criteria:

* A history of coronary artery disease, heart failure, stroke, diabetes, malignancy, chronic pulmonary, kidney or rheumatologic disease, muscle pain/fatigue, smoking within the past 5 years, regular use of any medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2021-05-07 (Actual)

PRIMARY OUTCOMES:
Change in proportion of CD59 on the endothelial cell (EC) surface (the percent [%] of the total cellular CD59 protein that is expressed on the endothelial cell surface). | Up to 28 days
  Outcome 1 will be assessed before and after 4 weeks of atorvastatin or placebo. Each patient 28-day follow-up value will be compared with baseline value. There is no reference range for this marker of complement regulation. The percent of total CD59 located on the EC plasma membrane will be quantified using immunofluorescence and confocal microscopy. This is a single outcome measure. The unit is percent (%) of the total cellular CD59 protein that is expressed on the endothelial cell surface.

SECONDARY OUTCOMES:
MAC deposition on EC surface (measurement unit is fluorescent area quantified as micrometer square). | Up to 28 days
  Outcome 2 will be assessed before and after 4 weeks of atorvastatin or placebo. Each patient 28-day follow-up value will be compared with baseline value. This is a single outcome measure. There is no reference range for this marker of complement regulation. MAC deposition on the EC plasma membrane will be quantified using immunofluorescence and confocal microscopy and expressed as the fluorescent area in micrometer square.
ORP1L (late endosome protein) and VAPB (endoplasmic reticulum protein) interaction (measurement unit is fluorescent area quantified as micrometer square). | 1 day
  Outcome 3 will be assessed at baseline between healthy control and OSA group and baseline vs post CPAP in OSA patients.

OTHER OUTCOMES:
Derlin and VAPB interaction | 1 day
  healthy controls vs OSA patients and baseline vs post CPAP in OSA patients
Lipid droplets in endothelial cells | 1 day
  healthy controls vs OSA patients
free cholesterol content in endothelial cells | 1 day
  healthy controls vs OSA patients
ABCA1 and G1 mRNA expression in endothelial cells | 1 day
  healthy controls vs OSA patients
ER stress markers mRNA expression in endothelial cells | 1 day
  healthy controls vs OSA patients

CONTACTS AND LOCATIONS:
Overall Officials: Sanja Jelic, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shah R, Patel N, Emin M, Celik Y, Jimenez A, Gao S, Garfinkel J, Wei Y, Jelic S. Statins Restore Endothelial Protection against Complement Activity in Obstructive Sleep Apnea: A Randomized Clinical Trial. Ann Am Thorac Soc. 2023 Jul;20(7):1029-1037. doi: 10.1513/AnnalsATS.202209-761OC. PMID 36912897